CLINICAL TRIAL: NCT00631150
Title: A Phase IV-Pharmacovigilance Study of Keppra Greece - S.K.A.T.E.: Safety of Keppra as Adjunctive Therapy in Epilepsy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Study Director, UCB
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N01035
Record Dates: First submitted 2008-02-27; First posted 2008-03-07 (Estimated); Last update posted 2013-11-15 (Estimated); Status verified 2009-09

CONDITIONS: Epilepsy
Keywords: Levetiracetam; Keppra
MeSH Terms: conditions — Epilepsy | interventions — Levetiracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Levetiracetam (Keppra)

SUMMARY:
Patients in community-based practices correspond to the 25% of patients who need a first add-on drug when not controlled by their standard monotherapy drug. This was a therapeutic use trial in which the population corresponds more closely to that seen in daily clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* partial onset seizures with or without secondary generalisation with epilepsy.

Exclusion Criteria:

* hypersensitivity to levetiracetam or other pyrrolidone derivatives or to any of the excipients.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2003-03; Primary Completion 2004-07 (Actual); Study Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
Safety and the tolerability of Keppra in a broad population of patients.

SECONDARY OUTCOMES:
Obtain further information about optimal daily dose.

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)